CLINICAL TRIAL: NCT03578718
Title: Evaluation of the Interest of a Specialist in Dermatology for Dermatopediatric Consultations
Acronym: HLSkinPed
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-A00088-47
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-06

CONDITIONS: Dermatologic Disease; Pediatric ALL; Collaboration
MeSH Terms: conditions — Skin Diseases; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Dermatologic diseases, of very different etiology and variable severity, represent a major motivation for consultation (in private consultations and in emergency departments), thus leading pediatricians to frequently turn to dermatologic advice.

The principal aim is to estimate the degree of concordance of the main diagnosis between a pediatrician and a pediatric dermatologist.

The secondary aims is to estimate the degree of concordance of the treatment, advices and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Under 18 years old
* consultating for dermatologic problem in emergency department (1 department) or private pediatric center (1 center)
* signed consent
* consécutives consultations

Exclusion Criteria:

* no consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: all patients Under 18 years old consulting for a dermatological problem in emergency department or in a private pediatric consultation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-06-25 (Estimated); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
principal diagnosis | baseline
  % of concordance between diagnosis (dermatologist/pediatric)

SECONDARY OUTCOMES:
treament | baseline
  % of concordance between treatment (dermatologist/pediatric)
advices | baseline
  % of concordance between advices(dermatologist/pediatric)
follow-up | baseline
  % of concordance between follow-up (dermatologist/pediatric)